CLINICAL TRIAL: NCT01619800
Title: The impAct of Blended Sensor Optimization on resoLVing Chronotropic Incompetence: ABSOLVE CI
Brief Title: The Effect of Blended Sensor Efficiency on Relieving the Heart's Inability to Increase Its Rate During Exercise
Acronym: ABSOLVE CI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to poor enrollment.
Sponsor: Vivek Reddy (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor Of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-02-333-05
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Chronotropic Incompetence
Keywords: Chronotropic Incompetence; Pacemaker; Mount Sinai School of Medicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blended Sensor Optimization (BSO) (Experimental): Patients in this arm will undergo pacemaker placement and will have blended sensor optimization. Minute Ventilation will be optimized/activated
  Interventions: Device: Blended Sensor Optimization (BSO)
- Accelerometer Alone (AA) (Sham Comparator): Patients in this arm will undergo pacemaker implantation but will not have Minute Ventilation Sensor activated. Only accelerometer will remain active
  Interventions: Device: Accelerometer Alone (AA)

INTERVENTIONS:
Device: Blended Sensor Optimization (BSO) — At wound check (POD#1 and 1 Week F/U), histograms from device interrogation obtained from patients in the BSO group are assessed, and these patients undergo optimization. A hall walk and stair climbing exercise will be performed and MV optimized using trending data to hit the following targets:
  HR at Rest: 60 HR upon slow walking: 100 HR upon brisk walking: 115-120 HR upon climbing stairs: 130-135 Patients will undergo optimization, and be instructed that their device may have been optimized.
  Arms: Blended Sensor Optimization (BSO)
Device: Accelerometer Alone (AA) — Patients in the AA group will also undergo device interrogation, and will perform a hall walk and stair climbing exercise. Afterwards, these patients will undergo a sham optimization by placing the PPM interrogation laptop device over there pacemaker, and instructing the patients that their device may have been optimized.
  Arms: Accelerometer Alone (AA)

SUMMARY:
The goal of this trial is to test the effect/benefit of a FDA approved blended pacemaker sensor which responds only by comparing physical activity, heart rate, and breathing rate; compared to the accelerometer pacemaker sensor which respond only by comparing physical activity and the heart rate in patients whose heart is unable increase its heart rate according to increase physical activity or demand (Chronotropic Incompetence). Only one pacemaker family will be used in this clinical trial whereas the "out of box" configuration is the blended sensor which can also be made to act only as an accelerometer.

DETAILED DESCRIPTION:
Objective: The goal of this trial is to test the impact of individualized blended sensor optimization on chronotropic response, compared with accelerometer use alone, in patients with chronotropic incompetence who are planned to undergo permanent pacemaker (PPM) implantation.

Study Population: The study population will consist of patients who suffer from the heart's inability to increase its heart rate according to increased physical activity or demand (chronotropic incompetence). These patients are planned to undergo permanent pacemaker (PPM) implantation.

PRIMARY ENDPOINT: Improvement in chronotropic competence as defined as an increase in age-predicted maximum heart rate (APMHR) which is defined as 220 beats per minute (bpm) minus patient's age in years. Age-predicted heart rate reserve (APMHR) defined as APMHR minus patient's heart rate at rest. Observe the maximal heart rate during exercise test with decrease in oxygen consumption at each stage and also at peak effort.

SECONDARY ENDPOINT:

1. Quality of life.
2. Procedural safety as defined by the number of complications within 1week associated with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Evidence of chronotropic incompetence on exercise or pharmacological stress test defined as the inability to achieve 85% or greater of Age-predicted heart rate reserve (APMHR)
* Legal status to give informed consent specific to state and national law.
* Planned for PPM implantation and meets current guidelines for PPM therapy.

Exclusion Criteria:

* Inability to give informed consent
* Inability to comply with the follow-up visit schedule.
* Unable to participate in stress testing (exercise or pharmacological).
* Previous PPM implantation
* A life expectancy of less than 12 months per physician discretion
* Enrolled in any concurrent study, without Boston Scientific written approval.
* Pregnancy
* Unstable chest pain
* Stroke within 30 days
* Heart attack within 90 days
* Stress Test Exclusion Criteria: No evidence of Chronotropic incompetence on exercise or pharmacological stress test, defined as the ability to achieve 85% or greater of APMHR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blended Sensor Optimization (BSO) | Accelerometer Alone (AA)
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — study terminated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blended Sensor Optimization (BSO) | Accelerometer Alone (AA) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Changed in Stress Test at 6 Months as Compared to Baseline
Description: An Exercise or Dobumatime Stress Test to be performed to assess primary outcome measure.
Time Frame: baseline and 6 months
Arm/Group | Blended Sensor Optimization (BSO) | Accelerometer Alone (AA)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Blended Sensor Optimization (BSO) | Accelerometer Alone (AA)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
2 subjects enrolled, unable to meet goal of 38 enrollments. Data not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes